CLINICAL TRIAL: NCT05793567
Title: Assessment of Microcirculatory Function in Type 2 Myocardial Infarction
Brief Title: A Study of Microcirculatory Function in Type 2 Myocardial Infarction (T2MI)
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Claire E. Raphael, Principal Investigator, Mayo Clinic
Other Study IDs: 22-012721
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction; Coronary Microvascular Disease
MeSH Terms: conditions — Myocardial Infarction; Microvascular Angina | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- T2MI Patients: Patients with T2MI and no epicardial coronary stenosis >50% will be prospectively enrolled and undergo a routine standard of care coronary angiogram with coronary reactivity testing (CRT).
  Interventions: Diagnostic Test: Coronary angiogram with coronary reactivity testing (CRT)
- Controls: Patients with atypical chest pain and no obstructive disease on coronary angiogram who have been referred for investigation of suspected CMD and have a clinical indication for CMD testing will be retrospectively enrolled and data collected from a previous routine standard of care coronary angiogram with coronary reactivity testing (CRT) will be utilized.

INTERVENTIONS:
Diagnostic Test: Coronary angiogram with coronary reactivity testing (CRT) — CRT is an angiography procedure (using X-ray) to examine the small blood vessels in the heart and how they respond to three drugs (adenosine, acetylcholine and nitroglycerin) as per clinical protocol.
  Groups: T2MI Patients

SUMMARY:
The purpose of this research is to find out if patients with Type 2 Myocardial Infarction (T2MI) without significant epicardial coronary artery disease (CAD) have a greater chance of having coronary microvascular disease (CMD).

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Structurally normal heart (normal LV and RV function, no more than mild valvular heart disease)
* For controls: atypical chest pain with indication for CMD testing
* For T2MI: meet criteria for T2MI according to the 4th Universal definition of MI (rise/fall of troponin with at least 1 value >99th centile+ evidence of symptoms or signs of myocardial ischemia)

Exclusion Criteria:

* Acute coronary event (evidence of plaque rupture, fissure or dissection on coronary angiogram)
* Known to have angiographically significant CAD/pressure wire positive for epicardial CAD
* Inability to receive heparin products
* Allergy/contraindication to acetylcholine/adenosine/nitroglycerine products
* Prior coronary artery bypass grafting
* Pregnancy (if sexually active woman of reproductive age, need negative pregnancy test prior to proceeding with coronary angiography - this is standard of care in cath lab)
* Asthma with prior ICU admission due to bronchospasm/need for invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects receiving care at Mayo Clinic in Rochester, MN identified with T2MI and controls with atypical chest pain with indication for CMD testing will be enrolled in this study. Both groups will have no epicardial coronary stenosis >50% or obstructive disease.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Coronary Flow Reserve (CFR) | Baseline
  The CFR will be calculated as a ratio of coronary flow at peak hyperemia /coronary flow at rest.

SECONDARY OUTCOMES:
Backward Compression Wave (BCW) | Baseline
  The BCW is a measure of increased microvascular resistance during systole.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Raphael, MBBS, PhD., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials